CLINICAL TRIAL: NCT04699448
Title: Genetic Predisposition and Body Weight Regulation. Evaluation of Target-genes in Overweight and Obese Adults, Under Different Dietary Interventions.
Brief Title: Gene-diet Interactions on Body Weight Regulation and Lifestyle Parameters.
Acronym: iMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, GEORGIOS DEDOUSSIS, Professor of Molecular Genetics - Nutrigenetics, Vice Rector of Academic of Affairs and Quality Assurance, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1800/13-06-2019
Record Dates: First submitted 2020-12-18; First posted 2021-01-07 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Gene-diet Interactions; Overweight and Obesity; Body Weight Changes; Health Status; Quality of Life
Keywords: Gene-diet interactions; Nutritional Intervention; Online Self-assessment Tools; Body Composition; Lifestyle characteristics
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-protein hypocaloric diet (Active Comparator): Composition of hypocaloric diet: protein:40%,carbohydrates:30% and fat:30%.
  Interventions: Other: Nutritional intervention.
- High-carbohydrate hypocaloric diet (Active Comparator): Composition of hypocaloric diet: carbohydrate 60%, protein:18% and fat:22%
  Interventions: Other: Nutritional intervention.

INTERVENTIONS:
Other: Nutritional intervention. — Diets designed for body weight loss, based on different macronutrient content.

SUMMARY:
Increased body weight leading to the development and the establishment of overweight and obesity, has a growing detrimental effect on overall health status and quality of life. Latest research has been focusing on the direct influence of dietary habits on body weight regulation and its synergistic effect with genetic predisposition. The synergistic effect of genetic makeup and dietary habits constitute a major contributing factor, specifically in its manifestation on parameters of the cardiometabolic profile of individuals with elevated body weight.

In this context, the aim of the present study is to investigate the effect of two hypocaloric diets with different macronutrient content (a high-carbohydrate/low-fat and a high-protein one) on the body weight loss of an overweight and/or obese adult, Greek population. Moreover, the study aims to explore gene-diet interactions between obesity and weight loss- related target genes and adherence to the proposed dietary schemes. It will further examine influences of the aforementioned factors on body composition, anthropometric indices, such as waist circumference, biochemical biomarkers related to cardiometabolic control and parameters of lifestyle, such as sleep quality.

More specifically, 300 participants will be allocated into two groups, following either the high-carbohydrate/low-fat diet or the high-protein diet, for a duration of 3 months. Volunteers will participate in in-person meetings, at baseline and at three months after the beginning of the intervention. Anthropometric measurements and collection of blood samples will take place in each meeting. Demographic data and data on family and medical history, dietary habits, adherence to the Mediterranean diet, overall health status and physical activity will be collected at baseline. Participants will be provided with nutritional counselling and support both at the beginning and throughout the intervention. Participants will further report their monthly progress by completing online questionnaires (namely concerning their body weight, overall health status, physical activity and sleep quality), via use of an online assessment tool developed by our team.

The effect of the intervention will be evaluated using anthropometric indices, body composition markers and biochemical biomarkers of cardiometabolic control, pre- and post- intervention. Gene-diet interactions will be assessed via genotyping of DNA samples and statistical analyses will take place via statistical packages, such as PLINK v.1.9.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 18 to 65 years of age.
* Body Mass Index of over 25kg/m2 (presence of overweight or obesity)

Exclusion Criteria:

* Pregnancy or lactation.
* Unregulated comorbidities (i.e. type 1 or 2 diabetes, cardiovascular disease, gastrointestinal disorders, mental illness, dietary disorders)
* Dietary supplements aiming at body weight loss
* Parallel participation in a different research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Body Weight | 3 months
  Changes in body weight compared to baseline.

SECONDARY OUTCOMES:
Body fat percentage | 3 months
  Changes in body fat percentage compared to baseline.
Waist circumference | 3 months
  Changes in waist circumference compared to baseline.
Visceral fat | 3 months
  Changes in visceral fat compared to baseline.
Biochemical profile | 3 months
  Changes in biochemical biomarkers related to metabolic syndrome and cardiovascular disease risk (i.e. total cholesterol, glucose, triglyceride and HDL levels) compared to baseline.
Sleep quality | 3 months
  Changes in sleep quality characteristics compared to baseline. Assessment will take place via use of validated questionnaire.
Overall health status | 3 months
  Changes in the overall health status compared to baseline. Assessment will take place via use of validated questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Harokopio University, Athens, Kallithea, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray GA, Krauss RM, Sacks FM, Qi L. Lessons Learned from the POUNDS Lost Study: Genetic, Metabolic, and Behavioral Factors Affecting Changes in Body Weight, Body Composition, and Cardiometabolic Risk. Curr Obes Rep. 2019 Sep;8(3):262-283. doi: 10.1007/s13679-019-00353-1. PMID 31214942
- [Background] Shungin D, Winkler TW, Croteau-Chonka DC, Ferreira T, Locke AE, Magi R, Strawbridge RJ, Pers TH, Fischer K, Justice AE, Workalemahu T, Wu JMW, Buchkovich ML, Heard-Costa NL, Roman TS, Drong AW, Song C, Gustafsson S, Day FR, Esko T, Fall T, Kutalik Z, Luan J, Randall JC, Scherag A, Vedantam S, Wood AR, Chen J, Fehrmann R, Karjalainen J, Kahali B, Liu CT, Schmidt EM, Absher D, Amin N, Anderson D, Beekman M, Bragg-Gresham JL, Buyske S, Demirkan A, Ehret GB, Feitosa MF, Goel A, Jackson AU, Johnson T, Kleber ME, Kristiansson K, Mangino M, Leach IM, Medina-Gomez C, Palmer CD, Pasko D, Pechlivanis S, Peters MJ, Prokopenko I, Stancakova A, Sung YJ, Tanaka T, Teumer A, Van Vliet-Ostaptchouk JV, Yengo L, Zhang W, Albrecht E, Arnlov J, Arscott GM, Bandinelli S, Barrett A, Bellis C, Bennett AJ, Berne C, Bluher M, Bohringer S, Bonnet F, Bottcher Y, Bruinenberg M, Carba DB, Caspersen IH, Clarke R, Daw EW, Deelen J, Deelman E, Delgado G, Doney AS, Eklund N, Erdos MR, Estrada K, Eury E, Friedrich N, Garcia ME, Giedraitis V, Gigante B, Go AS, Golay A, Grallert H, Grammer TB, Grassler J, Grewal J, Groves CJ, Haller T, Hallmans G, Hartman CA, Hassinen M, Hayward C, Heikkila K, Herzig KH, Helmer Q, Hillege HL, Holmen O, Hunt SC, Isaacs A, Ittermann T, James AL, Johansson I, Juliusdottir T, Kalafati IP, Kinnunen L, Koenig W, Kooner IK, Kratzer W, Lamina C, Leander K, Lee NR, Lichtner P, Lind L, Lindstrom J, Lobbens S, Lorentzon M, Mach F, Magnusson PK, Mahajan A, McArdle WL, Menni C, Merger S, Mihailov E, Milani L, Mills R, Moayyeri A, Monda KL, Mooijaart SP, Muhleisen TW, Mulas A, Muller G, Muller-Nurasyid M, Nagaraja R, Nalls MA, Narisu N, Glorioso N, Nolte IM, Olden M, Rayner NW, Renstrom F, Ried JS, Robertson NR, Rose LM, Sanna S, Scharnagl H, Scholtens S, Sennblad B, Seufferlein T, Sitlani CM, Smith AV, Stirrups K, Stringham HM, Sundstrom J, Swertz MA, Swift AJ, Syvanen AC, Tayo BO, Thorand B, Thorleifsson G, Tomaschitz A, Troffa C, van Oort FV, Verweij N, Vonk JM, Waite LL, Wennauer R, Wilsgaard T, Wojczynski MK, Wong A, Zhang Q, Zhao JH, Brennan EP, Choi M, Eriksson P, Folkersen L, Franco-Cereceda A, Gharavi AG, Hedman AK, Hivert MF, Huang J, Kanoni S, Karpe F, Keildson S, Kiryluk K, Liang L, Lifton RP, Ma B, McKnight AJ, McPherson R, Metspalu A, Min JL, Moffatt MF, Montgomery GW, Murabito JM, Nicholson G, Nyholt DR, Olsson C, Perry JR, Reinmaa E, Salem RM, Sandholm N, Schadt EE, Scott RA, Stolk L, Vallejo EE, Westra HJ, Zondervan KT; ADIPOGen Consortium; CARDIOGRAMplusC4D Consortium; CKDGen Consortium; GEFOS Consortium; GENIE Consortium; GLGC; ICBP; International Endogene Consortium; LifeLines Cohort Study; MAGIC Investigators; MuTHER Consortium; PAGE Consortium; ReproGen Consortium; Amouyel P, Arveiler D, Bakker SJ, Beilby J, Bergman RN, Blangero J, Brown MJ, Burnier M, Campbell H, Chakravarti A, Chines PS, Claudi-Boehm S, Collins FS, Crawford DC, Danesh J, de Faire U, de Geus EJ, Dorr M, Erbel R, Eriksson JG, Farrall M, Ferrannini E, Ferrieres J, Forouhi NG, Forrester T, Franco OH, Gansevoort RT, Gieger C, Gudnason V, Haiman CA, Harris TB, Hattersley AT, Heliovaara M, Hicks AA, Hingorani AD, Hoffmann W, Hofman A, Homuth G, Humphries SE, Hypponen E, Illig T, Jarvelin MR, Johansen B, Jousilahti P, Jula AM, Kaprio J, Kee F, Keinanen-Kiukaanniemi SM, Kooner JS, Kooperberg C, Kovacs P, Kraja AT, Kumari M, Kuulasmaa K, Kuusisto J, Lakka TA, Langenberg C, Le Marchand L, Lehtimaki T, Lyssenko V, Mannisto S, Marette A, Matise TC, McKenzie CA, McKnight B, Musk AW, Mohlenkamp S, Morris AD, Nelis M, Ohlsson C, Oldehinkel AJ, Ong KK, Palmer LJ, Penninx BW, Peters A, Pramstaller PP, Raitakari OT, Rankinen T, Rao DC, Rice TK, Ridker PM, Ritchie MD, Rudan I, Salomaa V, Samani NJ, Saramies J, Sarzynski MA, Schwarz PE, Shuldiner AR, Staessen JA, Steinthorsdottir V, Stolk RP, Strauch K, Tonjes A, Tremblay A, Tremoli E, Vohl MC, Volker U, Vollenweider P, Wilson JF, Witteman JC, Adair LS, Bochud M, Boehm BO, Bornstein SR, Bouchard C, Cauchi S, Caulfield MJ, Chambers JC, Chasman DI, Cooper RS, Dedoussis G, Ferrucci L, Froguel P, Grabe HJ, Hamsten A, Hui J, Hveem K, Jockel KH, Kivimaki M, Kuh D, Laakso M, Liu Y, Marz W, Munroe PB, Njolstad I, Oostra BA, Palmer CN, Pedersen NL, Perola M, Perusse L, Peters U, Power C, Quertermous T, Rauramaa R, Rivadeneira F, Saaristo TE, Saleheen D, Sinisalo J, Slagboom PE, Snieder H, Spector TD, Stefansson K, Stumvoll M, Tuomilehto J, Uitterlinden AG, Uusitupa M, van der Harst P, Veronesi G, Walker M, Wareham NJ, Watkins H, Wichmann HE, Abecasis GR, Assimes TL, Berndt SI, Boehnke M, Borecki IB, Deloukas P, Franke L, Frayling TM, Groop LC, Hunter DJ, Kaplan RC, O'Connell JR, Qi L, Schlessinger D, Strachan DP, Thorsteinsdottir U, van Duijn CM, Willer CJ, Visscher PM, Yang J, Hirschhorn JN, Zillikens MC, McCarthy MI, Speliotes EK, North KE, Fox CS, Barroso I, Franks PW, Ingelsson E, Heid IM, Loos RJ, Cupples LA, Morris AP, Lindgren CM, Mohlke KL. New genetic loci link adipose and insulin biology to body fat distribution. Nature. 2015 Feb 12;518(7538):187-196. doi: 10.1038/nature14132. PMID 25673412